CLINICAL TRIAL: NCT04440436
Title: Phase I/II Clinical Study to Evaluate the Safety and Efficacy of IM19 Chimeric Antigen Receptor T Cells(CAR-T) in the Treatment of Recurrent or Refractory (R/R) CD19 Positive Aggressive Non-Hodgkin's Lymphoma
Brief Title: Assessment of Safety and Efficacy of IM19 for Recurrent or Refractory (R/R) Non-Hodgkin's Lymphoma(NHL) Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Collaborators: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SD45
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: NHL
MeSH Terms: interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IM19 CAR-T cells (Experimental): IM19 CAR-T cells be administrated in two dose level
  Interventions: Drug: IM19 CAR-T Cells

INTERVENTIONS:
Drug: IM19 CAR-T Cells — IM19 CAR-T cells
  Drug: Fludarabine
  Two days before cell infusion, all patients will be treated with fludarabine for 3 days
  Drug: Cyclophosphamide
  Two days before cell infusion, all patients will be treated with Cyclophosphamide for 3 days
  Other Names: Fludarabine; Cyclophosphamide

SUMMARY:
This is a phase I/II, multicenter study to assess the efficacy and safety of IM19 CAR-T cells in adult with R/R Non-Hodgkins Lymphoma in China.

DETAILED DESCRIPTION:
This is a phase Ⅰ/Ⅱ. The phase I is a single-center study. The main objective is to evaluate the safety of IM19 CAR-T cell therapy for patients with relapsed or refractory CD19-positive invasion of non-Hodgkin's lymphoma. The phase Ⅱ is a multi-center study,The main goal is to evaluate the efficacy of IM19 CAR-T cells in the treatment of patients with relapsed or refractory CD19-positive invasion of non-Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with relapsed or refractory invasive non-Hodgkin's lymphoma, confirmed by CD19 positive cytology or histology, specific types.
* CD20 positive patients undergo corresponding targeted therapy.
* Patients must have evaluable evidence of disease (according to Lugano 2014 standards).
* ≥ 18 years old.
* The expected survival period is more than 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Women of childbearing age have a negative blood pregnancy test before the start of the trial and agree to have effective contraceptive measures during the trial until the last follow-up
* Participate voluntarily in this experiment and sign the informed consent.

Exclusion Criteria:

* The investigators judged patients with gastrointestinal lymph nodes and/or central nervous system involvement who may be at risk for CAR-T treatment.
* Subject has graft-versus-host reactions and need to use immunosuppressants; or suffer from autoimmune disease
* Subject has used chemotherapy or radiotherapy within three days before the blood collection period.
* Subject has used systemic steroid drugs within 5 days before the blood collection period (except for recent or current inhaled steroids).
* Those who use drugs that stimulate bone marrow hematopoietic cells to produce drugs within 5 days before the blood collection
* Subject has used any gene therapy products before.
* Subject with a history of epilepsy or other central nervous system diseases.
* Active Hepatitis B Virus or Hepatitis C Virus infections
* The subject with other tumors in the past 5 years.
* Within 14 days before enrollment, there was active infection or uncontrollable infection requiring systemic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-06-04 (Actual); Primary Completion 2022-06-04 (Estimated); Study Completion 2035-06-04 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) at 90 days | 90 days
  The primary endpoint was ORR 90 days after IM19 infusion

CONTACTS AND LOCATIONS:
Overall Officials: Yuqin Song, MD, PhD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No